CLINICAL TRIAL: NCT00290251
Title: Evaluation of Whether the Selective Progesterone Receptor Modulator CDB-2914 Can Shrink Leiomyomata
Brief Title: Treatment of Uterine Fibroids With the Selective Progesterone Receptor Modulator CDB-2914
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: HRA Pharma (Industry)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 060090; 1ZIAHD000637-17 (NIH); 06-CH-0090 (Other: NIH IRB)
Record Dates: First submitted 2006-02-10; First posted 2006-02-10 (Estimated); Results first posted 2012-12-18 (Estimated); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Leiomyoma
Keywords: Endometrium; Progesterone; Estrogen; Fibroid; Hysterectomy; Leiomyoma; Uterine Fibroids; Fibroids
MeSH Terms: conditions — Leiomyoma | interventions — ulipristal acetate; ulipristal

STUDY DESIGN:
Intervention Model Description: Subjects were studied during a single baseline menstrual cycle followed by a cross-over into three arms (active treatment at one of two doses, or placebo) given for three menstrual cycles
Who Masked: Participant, Investigator
Masking Description: study agents were formulated in identical looking capsules
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- ulipristal acetate -20 mg (Active Comparator): 20 mg daily dose ulipristal acetate for three menstrual cycles or up to 102 days
  Interventions: Drug: ulipristal acetate 20 mg
- ulipristal acetate - 10 mg (Active Comparator): 10 mg daily dose ulipristal acetate for three menstrual cycles or up to 102 days
  Interventions: Drug: ulipristal acetate 10 mg
- Placebo (Placebo Comparator): Placebo taken daily for three menstrual cycles or up to 102 days
  Interventions: Drug: placebo
- Pre-ulipristal acetate 10 mg (No Intervention): Subjects were studied during one baseline cycle without any intervention before entering ulipristal acetate 10 mg arm
- Pre-ulipristal acetate 20 mg (No Intervention): Subjects were studied during one baseline cycle without any intervention before entering ulipristal acetate 20 mg arm
- Pre-placebo (No Intervention): Subjects were studied during one baseline cycle without any intervention before entering placebo arm

INTERVENTIONS:
Drug: ulipristal acetate 20 mg — ulipristal acetate at a daily dose of 20 mg, given once daily for three menstrual cycles or 90 - 102 days if amenorrheic
  Other Names: VA2914; CDB-2914
  Arms: ulipristal acetate -20 mg
Drug: ulipristal acetate 10 mg — 10 mg given daily for three menstrual cycles or 90 - 102 days
  Other Names: VA2914; CDB2914
  Arms: ulipristal acetate - 10 mg
Drug: placebo — placebo given once daily for 3 menstrual cycles or 90 - 102 days
  Arms: Placebo

SUMMARY:
This study will evaluate whether the experimental drug ulipristal acetate can shrink uterine fibroids in pre-menopausal women.

DETAILED DESCRIPTION:
Uterine leiomyomata (fibroids) are a common benign tumor of the uterine muscle in pre-menopausal women that may cause bleeding, pelvic pain and pressure. Because fibroids grow in the presence of estrogen, medical therapies that decrease estrogen levels (like Gonadotropin releasing hormone,GnRH analog) cause fibroids to shrink and so may relieve symptoms. However, such medication can only be given short-term and has inconvenient side effects such as hot-flashes. Thus, many women with symptomatic fibroids choose to have them removed surgically, either individually or by removing the uterus via hysterectomy.

Women between 25 and 50 years of age who have regular menstrual cycles and a history of uterine fibroids that cause heavy bleeding, pressure, or pain may be eligible for this study. Candidates are screened with a medical history and physical examination, including breast and pelvic examination, blood and urine tests, a quality-of-life questionnaire, and a home urine test for leuteinizing hormone (LH) surge. They are given a diary to record the LH surge, days of vaginal spotting or bleeding, and symptoms. Participation includes the following:

Baseline Studies (First Menstrual Cycle)

* Magnetic resonance imaging (MRI): The subject lies in the MRI scanner, a narrow cylinder with a strong magnetic field, for imaging the uterus.
* Saline hysterosonogram: This is an ultrasound examination of the uterus. A speculum is placed in the vagina and a small amount of liquid is inserted into the uterus. A probe is then inserted into the vagina. The probe emits and receives sound waves that are used to visualize the fibroids and surrounding structures.

Study Drug Phase (Second through Fourth Menstrual Cycles)

* Subjects are randomly assigned to take ulipristal acetate or placebo (inactive compound) once a day by mouth on an empty stomach for three menstrual cycles or up to 102 days if menstrual cycles are irregular or stop.
* Pregnancy test on first or second day of every menstrual cycle.
* Blood tests every 2 weeks to measure effects of study medication on hormones, blood count, blood chemistries and liver function.
* 24-hour urine collections three times during the study, about once a month, to measure cortisol and check adrenal gland function.
* Repeat transvaginal ultrasound after 4-6 weeks of study drug to check fibroid growth.
* Repeat hysterosonogram and MRI within 2 weeks of surgery to count and measure the fibroids. or placebo (inactive compound) once a day by mouth on an empty stomach for three menstrual cycles or up to 102 days if menstrual cycles are irregular or stop.
* Pregnancy test on first or second day of every menstrual cycle.
* Blood tests every 2 weeks to measure effects of study medication on hormones, blood count, blood chemistries and liver function.
* 24-hour urine collections three times during the study, about once a month, to measure cortisol and check adrenal gland function.
* Repeat transvaginal ultrasound after 4-6 weeks of study drug to check fibroid growth.
* Repeat hysterosonogram and MRI within 2 weeks of surgery to count and measure the fibroids. or placebo (inactive compound) once a day by mouth on an empty stomach for three menstrual cycles or up to 102 days if menstrual cycles are irregular or stop.
* Pregnancy test on first or second day of every menstrual cycle.
* Blood tests every 2 weeks to measure effects of study medication on hormones, blood count, blood chemistries and liver function.
* 24-hour urine collections three times during the study, about once a month, to measure cortisol and check adrenal gland function.
* Repeat transvaginal ultrasound after 4-6 weeks of study drug to check fibroid growth.
* Repeat hysterosonogram and MRI within 2 weeks of surgery to count and measure the fibroids.

ELIGIBILITY:
INCLUSION CRITERIA:

* Female gender-to evaluate effects in the target population for clinical trials.
* History of uterine leiomyoma causing symptoms of bleeding, pressure, or pain, as defined by the American College of Obstetrics and Gynecology (ACOG) practice bulletin:
* Excessive uterine bleeding will be evidenced by either of the following-profuse bleeding with flooding or clots or repetitive periods lasting for more than 8 days; or anemia due to acute or chronic blood loss;

OR

* Pelvic discomfort caused by leiomyomata, either acute and severe or chronic lower abdominal or low back pressure or bladder pressure with urinary frequency not due to urinary tract infection.
* Uterine leiomyoma(ta) of at least 2 cm size.
* In good health. Chronic medication use is acceptable except for glucocorticoid use. Other chronic medication use may be acceptable at the discretion of the research team. Interval use of over-the-counter drugs is acceptable but must be recorded.
* Menstrual cycles of 24 - 35 days.
* Hemoglobin greater than 10 g/dL (for those wishing surgery); iron may be administered to improve red blood cell counts.
* Willing and able to comply with study requirements.
* Age 25 to 50.
* Using mechanical (condoms, diaphragms) sterilization or abstinence methods of contraception for the duration of the study.
* Negative urine pregnancy test.
* Body mass index (BMI) less than or equal to 33, if a surgical candidate or less than or equal to 35, if not a surgical candidate.
* Creatinine less than 1.3 mg/dL.
* Liver function tests within 130% of upper limit.
* If interested in hysterectomy, no desire for fertility.

EXCLUSION CRITERIA:

* Significant abnormalities in the history, physical or laboratory examination.
* Pregnancy.
* Lactation.
* Use of oral, injectable or inhaled glucocorticoids or megestrol within the last year.
* Unexplained vaginal bleeding.
* History of malignancy within the past 5 years.
* Use of estrogen or progesterone-containing compounds, such as oral contraceptives and hormone replacement therapy, within 8 weeks of study entry, including transdermal, injectable, vaginal and oral preparations.
* Use of agents known to induce hepatic P450 enzymes; use of imidazoles.
* Current use of Gonadotropin-releasing hormone (GnRH) analogs or other compounds that affect menstrual cyclicity.
* Follicle stimulating hormone (FSH) greater than 20 IU/mL.
* Untreated cervical dysplasia.
* Need for interval use of narcotics.
* Abnormal adnexal/ovarian mass.
* Use of herbal medication having estrogenic or antiestrogenic effects within the past 3 months.
* Contradiction to anesthesia, for women planning surgery.
* Genetic causes of leiomyomata.
* Previous participation in the study.
* Known recent rapid growth of fibroids, defined as a doubling in size in six months.

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2006-02; Primary Completion 2009-07 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynnette K Nieman, MD, Principal Investigator — NICHD, NIH
Locations (2):
- United States (2):
  - NIH Clinical Center, Bethesda, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Batista MC, Cartledge TP, Zellmer AW, Merino MJ, Axiotis C, Loriaux DL, Nieman LK. Delayed endometrial maturation induced by daily administration of the antiprogestin RU 486: a potential new contraceptive strategy. Am J Obstet Gynecol. 1992 Jul;167(1):60-5. doi: 10.1016/s0002-9378(11)91627-5. PMID 1442957
- [Background] Burroughs KD, Howe SR, Okubo Y, Fuchs-Young R, LeRoith D, Walker CL. Dysregulation of IGF-I signaling in uterine leiomyoma. J Endocrinol. 2002 Jan;172(1):83-93. doi: 10.1677/joe.0.1720083. PMID 11786376
- [Background] Cadepond F, Ulmann A, Baulieu EE. RU486 (mifepristone): mechanisms of action and clinical uses. Annu Rev Med. 1997;48:129-56. doi: 10.1146/annurev.med.48.1.129. PMID 9046951
- [Background] Levens ED, Wesley R, Premkumar A, Blocker W, Nieman LK. Magnetic resonance imaging and transvaginal ultrasound for determining fibroid burden: implications for research and clinical care. Am J Obstet Gynecol. 2009 May;200(5):537.e1-7. doi: 10.1016/j.ajog.2008.12.037. Epub 2009 Mar 9. PMID 19268886
- [Background] Nieman LK, Blocker W, Nansel T, Mahoney S, Reynolds J, Blithe D, Wesley R, Armstrong A. Efficacy and tolerability of CDB-2914 treatment for symptomatic uterine fibroids: a randomized, double-blind, placebo-controlled, phase IIb study. Fertil Steril. 2011 Feb;95(2):767-72.e1-2. doi: 10.1016/j.fertnstert.2010.09.059. Epub 2010 Nov 5. PMID 21055739
- [Derived] Parikh TP, Malik M, Britten J, Aly JM, Pilgrim J, Catherino WH. Steroid hormones and hormone antagonists regulate the neural marker neurotrimin in uterine leiomyoma. Fertil Steril. 2020 Jan;113(1):176-186. doi: 10.1016/j.fertnstert.2019.08.090. PMID 32033718
- [Derived] Lewis TD, Malik M, Britten J, Parikh T, Cox J, Catherino WH. Ulipristal acetate decreases active TGF-beta3 and its canonical signaling in uterine leiomyoma via two novel mechanisms. Fertil Steril. 2019 Apr;111(4):806-815.e1. doi: 10.1016/j.fertnstert.2018.12.026. Epub 2019 Mar 11. PMID 30871768
- [Derived] Ng SSM, Jorge S, Malik M, Britten J, Su SC, Armstrong CR, Brennan JT, Chang S, Baig KM, Driggers PH, Segars JH. A-Kinase Anchoring Protein 13 (AKAP13) Augments Progesterone Signaling in Uterine Fibroid Cells. J Clin Endocrinol Metab. 2019 Mar 1;104(3):970-980. doi: 10.1210/jc.2018-01216. PMID 30239831
- [Derived] Levens ED, Potlog-Nahari C, Armstrong AY, Wesley R, Premkumar A, Blithe DL, Blocker W, Nieman LK. CDB-2914 for uterine leiomyomata treatment: a randomized controlled trial. Obstet Gynecol. 2008 May;111(5):1129-36. doi: 10.1097/AOG.0b013e3181705d0e. PMID 18448745
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/B_2006-CH-0090.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Seventy-two women were screened for eligibility before being randomized to treatment. Of these only 42 were eligible to continue in the study.
Groups:
- Pre-ulipristal Acetate - 20 mg; Pre-ulipristal Acetate 10 mg: Women received no intervention for one menstrual cycle before entering ulipristal acetate 20 mg group
- Pre-placebo: Women received no intervention for one menstrual cycle before entering placebo group
- Ulipristal Acetate - 20 mg: Women received ulipristal acetate 20 mg/d
- Ulipristal Acetate- 10 mg: Women received ulipristal acetate at a daily dose of 10 mg for 90 - 102 days or three menstrual cycles.
- Placebo (PLC): Women received placebo capsules for 90 - 102 days or three menstrual cycles.
Period: Baseline (Month 1)
Arm/Group | Pre-ulipristal Acetate - 20 mg | Pre-ulipristal Acetate 10 mg | Pre-placebo | Ulipristal Acetate - 20 mg | Ulipristal Acetate- 10 mg | Placebo (PLC)
Started | 14 | 14 | 14 | 0 | 0 | 0
Completed | 14 | 14 | 14 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment 1 (Months 2-4)
Arm/Group | Pre-ulipristal Acetate - 20 mg | Pre-ulipristal Acetate 10 mg | Pre-placebo | Ulipristal Acetate - 20 mg | Ulipristal Acetate- 10 mg | Placebo (PLC)
Started | 0 (Subjects crossed over from no intervention baseline to treatment assignment) | 0 (Subjects crossed over from no intervention baseline to treatment assignment) | 0 (Subjects crossed over from no intervention baseline to treatment assignment) | 14 (Subjects crossed over from no intervention baseline to treatment assignment) | 14 (Subjects crossed over from no intervention baseline to treatment assignment) | 14 (Subjects crossed over from no intervention baseline to treatment assignment)
Completed | 0 | 0 | 0 | 13 | 13 | 12
Not Completed | 0 | 0 | 0 | 1 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 2
Not completed — headache | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Out of body experience | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: All women who received placebo
- Ulipristal Acetate 10 mg; Ulipristal Acetate 20 mg: All women who received Ulipristal Acetate - 20 mg
- Total: Total of all reporting groups
Arm/Group | Placebo | Ulipristal Acetate 10 mg | Ulipristal Acetate 20 mg | Total
Number analyzed (Participants) | 14 | 14 | 14 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 14 | 42
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 14 | 42
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 14 | 42

OUTCOME MEASURES:

1. Primary Outcome: Shrinkage of Fibroids - Size of Fibroids
Description: The primary outcome, fibroid volume, was calculated by an ellipsoid formula (π/6xd1xd2xd3) using orthogonal three-dimensional measurements taken from pelvic MRI scan. Individual volumes were summed to assess total fibroid volume for each woman, which were log-transformed before analysis. Women with paired MRI results were included in this intent to treat analysis, even if they did not take all study medication. Fibroids were included if they were seen on both studies.The absolute change in cm3 between baseline and end of treatment was calculated and its log was used for statistics and reporting the results in the data table below.
Time Frame: 3 months (baseline to end of treatment)
Population: Per protocol, including women with two MRIs regardless of whether they took all study medication. The two ulipristal acetate arms, 10 mg and 20 mg, were not different from each other (see statistical analysis 1) so they were combined for analysis of outcomes (in statistical analysis 2).
Measure: Mean (Standard Error); unit: logcm3
Groups:
- Ulipristal Acetate -20mg: Women received ulipristal acetate at 20 mg/day for 90 - 102 days or three menstrual cycles.
- Ulipristal Acetate - 10 mg: Women received ulipristal acetate at 10 mg/day for 90 - 102 days or three menstrual cycles.
- Placebo: Women received placebo capsules for 90 - 102 days or three menstrual cycles.
Arm/Group | Ulipristal Acetate -20mg | Ulipristal Acetate - 10 mg | Placebo
Number analyzed (Participants) | 13 | 13 | 12
logcm3 | -0.27 (0.07) | -0.18 (0.08) | 0.07 (0.78)
Statistical Analysis 1: Comparison: Ulipristal Acetate -20mg vs Ulipristal Acetate - 10 mg; Test type: Superiority; p = 0.43, t-test, 2 sided; performed on log-transformed delta change in total fibroid volume from baseline to end of treatment
Statistical Analysis 2: Comparison: Ulipristal Acetate -20mg vs Ulipristal Acetate - 10 mg vs Placebo; Ulipristal acetate groups one and two were first compared and found to be similar (see statistical analysis 1), so they were combined into a single treatment group for comparison to placebo group; Test type: Superiority or Other; p = 0.003, ANOVA; Performed on log-transformed delta change

2. Secondary Outcome: Short Form-36 and Uterine Fibroid Symptom Quality of Life
Description: The short form-36 (SF-36)and Uterine Fibroid Symptom Quality of Life (UFS-QOL) questionnaires were given before and at treatment end with scales of 0 - 100. SF-36 scales = mental and physical well-being. The UFS subscales are symptom severity, concern, activities, energy and mood, control, self-consciousness, sexual functioning compiled into an overall QOL score. Higher results indicate better QOL on all but symptom severity (higher = worse). The change in scores from baseline to end of treatment was calculated.
Time Frame: 3 months (Baseline to end of treatment 1)
Population: All completers received a questionnaire at the end of the three-month study. One woman in the placebo group did not complete the questionnaire. All women receiving ulipristal acetate were combined for analysis of QOL, to parallel the combined analysis done for the primary outcome measure.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Ulipristal Acetate -10 and 20mg: Women received ulipristal acetate at a daily dose of 10 or 20 mg for 90 - 102 days or three menstrual cycles.
Arm/Group | Ulipristal Acetate -10 and 20mg | Placebo
Number analyzed (Participants) | 26 | 11
units on a scale
  SF-36 Physical Component | 4.2 (1.2) | -1.5 (2.0)
  SF-36 Mental Component | 4.1 (1.5) | -2.2 (2.4)
  UFS Symptom Severity Score | -28.3 (4.2) | -4.2 (6.5)
  UFS Overall health related quality of life | 27.8 (3.6) | 8.6 (5.6)
  UFS Concern subscore | 46.1 (4.5) | 12.1 (6.9)
  UFS Energy/mood subscore | 19.2 (3.7) | 3.7 (5.8)
  UFS Control subscore | 20.3 (4.3) | 9.1 (6.8)
  UFS self-conscious subscore | 19.0 (4.7) | 15.8 (7.5)
  UFS sexual function subscore | 25.7 (5.5) | 18.7 (8.5)
  UFS activities subscore | 83.9 (4.4) | 56.1 (7.0)
  UFS composite bleeding subscore | 2.1 (0.2) | 0.4 (0.3)
Statistical Analysis 1: Comparison: Ulipristal Acetate -10 and 20mg vs Placebo; No sample size calculation was made; Test type: Superiority or Other; p < 0.05, ANOVA — The Delta of scores from treatment end to baseline was used to compare by ANOVA; Adjustment for age

ADVERSE EVENTS:
Time Frame: 120 - 132 days
Description: Women recorded specific adverse events on a calendar; there was also a write-in field. The number of women with at least one day of each symptom is reported.
Groups:
- Ulipristal Acetate -20mg: Women received ulipristal acetate at a daily dose of 20 mg for 90 - 102 days or three menstrual cycles.
- Pre-Ulipristal Acetate 20 mg: Women charted symptoms for one menstrual cycle before entering ulipristal acetate 20 mg group
- Pre-Ulipristal Acetate- 10 mg: Women charted symptoms for one menstrual cycle before entering ulipristal acetate 10 mg group
- Pre-Placebo: Women charted symptoms for one menstrual cycle before entering placebo group
Arm/Group | Ulipristal Acetate -20mg | Ulipristal Acetate- 10 mg | Placebo | Pre-Ulipristal Acetate 20 mg | Pre-Ulipristal Acetate- 10 mg | Pre-Placebo
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/14 | 0/14 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14 | 0/14 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 11/14 | 14/14 | 12/14 | 10/14 | 13/14 | 10/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ulipristal Acetate -20mg (N=14) | Ulipristal Acetate- 10 mg (N=14) | Placebo (N=14) | Pre-Ulipristal Acetate 20 mg (N=14) | Pre-Ulipristal Acetate- 10 mg (N=14) | Pre-Placebo (N=14)
Vaginal discharge (Reproductive system and breast disorders) | 6 (69) | 6 (50) | 4 (64) | 6 (21) | 3 (13) | 2 (8)
Nausea/vomiting (Gastrointestinal disorders) | 3 (4) | 2 (65) | 4 (10) | 0 (0) | 2 (2) | 1 (1) — Self-reported via calendar
Hot flashes (Skin and subcutaneous tissue disorders) | 5 (14) | 1 (64) | 1 (11) | 0 (0) | 0 (0) | 0 (0) — Self-reported via calendar
Non-menses Vaginal Bleeding (Reproductive system and breast disorders) | 3 (5) | 7 (107) | 3 (12) | 0 (0) | 2 (40) | 2 (7) — self-assessed via calendar
Breast pain (Reproductive system and breast disorders) | 6 (25) | 5 (95) | 8 (44) | 7 (20) | 3 (14) | 3 (10) — self-assessed via calendar
Abdominal pain (General disorders) | 10 (110) | 9 (37) | 10 (77) | 9 (29) | 11 (33) | 8 (32) — self-assessed via calendar
Pelvic pain (General disorders) | 5 (16) | 7 (16) | 5 (23) | 7 (23) | 5 (12) | 2 (14) — Self-assessed via calendar
Fatigue (General disorders) | 6 (25) | 8 (195) | 6 (75) | 9 (31) | 10 (76) | 6 (40) — self-assessed via calendar
Decreased appetitie (Gastrointestinal disorders) | 1 (4) | 1 (4) | 2 (11) | 1 (1) | 0 (0) | 2 (7) — self-assessed via calendar
Diarrhea (Gastrointestinal disorders) | 1 (4) | 3 (16) | 1 (5) | 2 (2) | 1 (2) | 0 (0) — self-assessed via calendar
Joint Pain (Musculoskeletal and connective tissue disorders) | 4 (33) | 1 (17) | 4 (40) | 5 (10) | 1 (1) | 3 (11) — self-assessed via calendar
Calf or Thigh pain (Musculoskeletal and connective tissue disorders) | 4 (32) | 1 (6) | 4 (19) | 4 (4) | 1 (3) | 1 (6) — self-assessed via calendar
Headache (General disorders) | 5 (13) | 7 (36) | 4 (24) | 2 (5) | 1 (2) | 2 (2) — self-assessed via calendar
Abdominal cramps (General disorders) | 2 (25) | 2 (9) | 3 (5) | 1 (4) | 1 (3) | 2 (6) — self-assessed via calendar
Mood changes (Psychiatric disorders) | 2 (3) | 0 (0) | 4 (16) | 1 (2) | 0 (0) | 1 (4) — self-assessed via calendar
Bloating (General disorders) | 0 (0) | 1 (4) | 1 (8) | 0 (0) | 0 (0) | 0 (0) — self-assessed via calendar
Leg swelling (General disorders) | 0 (0) | 1 (47) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — self-assessed via calendar and write-in option
Increased appetite (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 | 0 (0) | 0 (0) — self-assessed via calendar using write-in option
Back pain (Musculoskeletal and connective tissue disorders) | 4 (10) | 2 (15) | 2 (6) | 3 (20) | 2 (7) | 1 (5) — self-assessed by calendar
Depersonalization (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Out of body experience
Skin Rash (Skin and subcutaneous tissue disorders) | 1 (8) | 4 (43) | 2 (11) | 0 (0) | 0 (0) | 1 (6)
blood clots with menses (Reproductive system and breast disorders) | 1 (3) | 1 (5) | 3 (15) | 2 (8) | 0 (0) | 3 (6)
Lower extremity edema (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (76) | 0 (0)
constipaton (Gastrointestinal disorders) | 2 (6) | 0 (0) | 0 (0) | 2 (9) | 0 (0) | 0 (0)
weakness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
blurry vision (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
weight gain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hair loss (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
cold feet (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
galactorrhea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
food cravings (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
breast engorgement (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
disrupted sleep (Nervous system disorders) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less